CLINICAL TRIAL: NCT06363864
Title: Investigation of Metabolite Differences Between Taiwanese Metabolic Syndrome and Healthy Group Through Metabolomics
Brief Title: Investigation of Metabolomics Differences Between Metabolic Syndrome and Healthy Individuals in Taiwan
Status: Not yet recruiting | Type: Observational
Sponsor: Leeuwenhoek Laboratories Co. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: LL-IRB-2401
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy individuals
- Metabolic syndrome patients

SUMMARY:
The prevalence of metabolic syndrome in Taiwan has been increasing yearly. In this project, the database of blood test results from healthy and metabolic syndromes individuals will be analyzed to identify the small molecules related to the severity of metabolic syndrome. These identified small molecules could be used as biomarkers to predict the development of metabolic syndromes in the future.

ELIGIBILITY:
Inclusion Criteria:

* Capable adults weigh ≥ 50 kg

Exclusion Criteria:

* Not Taiwanese
* Having received oral antibiotics, immunosuppressants, and chemotherapy drugs in the past month
* Incapacity
* Limited disposing capacity
* Mental disorders or intellectual disabilities

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy individuals and patients with metabolic syndrom.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2024-04-14 (Estimated); Primary Completion 2029-10-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Concentration changes of small molecules in blood. | Up to six years
  Concentrations of small molecules in healthy individuals and metabolic syndrom patients will be analyzed to identify specific biomarkers for metabolic syndrome.